CLINICAL TRIAL: NCT06040788
Title: Effect of Tooth Angulation, Alveolar and Basal Bone Anatomical Characteristics on Soft and Hard Tissue Alterations Around Immediate Implants With Customized Healing Abutment. A 1-Year Randomized Clinical Trial
Brief Title: Effect of Tooth Angulation, Alveolar and Basal Bone Anatomical Characteristics on Soft and Hard Tissue Alterations Around Immediate Implants With Customized Healing Abutment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Lecturer in the department of Oral Medicine & Periodontology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDCE.N5
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Immediate Implant; Esthetic Zone; Customized Healing Abutment; Tissue Collapse; Tissue Dimensional Changes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immediate implant placement with customized healing abutment (Experimental)
  Interventions: Procedure: immediate implant placement with customized healing abutment

INTERVENTIONS:
Procedure: immediate implant placement with customized healing abutment — immediate implant placement with customized healing abutment

SUMMARY:
The goal of this clinical trial is to investigate the effect of different anatomical variations in terms of root angulation, alveolar bone and basal bone morphology on soft and hard tissue alterations in patients with non-restorable teeth in the inter-canine region undergoing immediate implantation. The main question it aims to answer are:

* Will the amount of collapse be greater when the root is proclined or outside the bone housing?
* Will no additional intervention be needed with immediate implants in the esthetic zone if we have better anatomy that will help hinder the collapse? Participants will receive immediate dental implants with customized healing abutments

ELIGIBILITY:
Inclusion Criteria:

Patient-related criteria:

* Adults at or above the age of 21.
* Non-restorable maxillary inter-canine tooth requiring extraction and needed an implant placing therapy.
* The failing tooth will have adjacent and opposing natural teeth.
* Sufficient mesial-distal and interocclusal space for placement of the implant and definitive restoration.
* Able to tolerate surgical periodontal procedures.
* Good oral hygiene.
* Compliance with the maintenance program.
* Provide informed consent.
* Accepts the one-year follow-up period.

Teeth related criteria:

* Intact thick biotype gingival tissue with at least 2mm band of keratinized tissue.
* Intact socket wall before the extraction, buccal bone thickness ≤1mm assessed by CBCT.
* Sufficient apical bone to place an immediate implant with minimum primary stability of 30Ncm.

Exclusion criteria:

* Patients diagnosed with periodontal diseases.
* Current or previous smokers.
* Pregnant and lactating females.
* Patients with medical conditions that would compromise the surgical procedures; uncontrolled diabetes mellitus, taking IV Bis-phosphonates for treatment of osteoporosis.
* Patients with active infection related at the site of implant/bone graft placement.
* Patients with parafunctional habits

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Amount of labiopalatal ridge collapse | 1 year
  radiographic Labiopalatal ridge collapse via CBCT
Amount of bone labial to the implant | 1 year
  Amount of bone labial to the implant at three levels 0, 2, and 5mmm below the alveolar crest via CBCT

SECONDARY OUTCOMES:
Amount of vertical crestal bone resorption in millimeters | 1 year
  Vertical crestal bone changes via CBCT in mm
Amount of change in buccal soft issue contour in mm3 | 1 year
  volumetric analysis of the amount of change in buccal soft issue contour in mm3
amount of Mid facial recession in millimeters | 1 year
  Mid facial recession in n millimeters
Pink esthetic score | 1 year
  1-14 scale